CLINICAL TRIAL: NCT01354093
Title: Utah Center for the Collaborative Study of the Role of the Macular Pigment Carotenoids in the Pathogenesis and Treatment of MacTel
Brief Title: The Role of Macular Pigment Carotenoids in the Pathogenesis and Treatment of Macular Telangiectasia Type 2 (MacTel)
Status: Completed | Type: Observational
Sponsor: Paul S. Bernstein (Other)
Responsible Party: Sponsor-Investigator, Paul S. Bernstein, Professor of Ophthalmology, University of Utah
Organization: University of Utah (Other)
Other Study IDs: 48834
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Idiopathic Juxtafoveal Telangiectasia
Keywords: MacTel; Macular telangiectasia type 2
MeSH Terms: conditions — Idiopathic Juxtafoveal Retinal Telangiectasia | interventions — Zeaxanthins

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MacTel Type 2 20 mg/day dose group: Participants will have macular telangiectasis type 2 as confirmed by the reading center. Participants will take 20 mg of zeaxanthin per day.
  Interventions: Drug: zeaxanthin
- MacTel Type 2 10 mg/day dose group: Participants will have macular telangiectasia type 2 as confirmed by the reading center. Participants will take 10 mg of zeaxanthin per day.
  Interventions: Drug: zeaxanthin

INTERVENTIONS:
Drug: zeaxanthin — 10 mg of EyePromise 10 (zeaxanthin) supplement, taken twice a day
  Groups: MacTel Type 2 20 mg/day dose group
Drug: zeaxanthin — 10 mg of EyePromise 10 (zeaxanthin) supplement, taken once a day
  Groups: MacTel Type 2 10 mg/day dose group

SUMMARY:
Macular telangiectasia type 2 ("MacTel Type 2") is an uncommon eye disorder that results in slow vision loss beginning in middle age. The macula is the central part of the retina, which lines the back of the eye like the film of a camera. The macula is responsible for central or reading vision. Telangiectasis refers to dilated, leaky vessels, for example varicose veins in the legs. One of the earliest manifestations of macular telangiectasia type 2 is an acquired reduction and/or redistribution of the macular pigment carotenoids at the foveal center. Currently, the biochemical mechanisms and clinical significance underlying these changes are not known, but it seems likely that better understanding of this phenomenon could lead to new interventions against MacTel.

The objectives of this study are to image the maculas of MacTel subjects using two-wavelength autofluorescence imaging and resonance Raman imaging to target the 7-degree radius pigment ring characteristic of macular telangiectasia type 2 in order to gain further insight into the significance of this early clinical sign, and to evaluate whether supplementation with oral zeaxanthin can normalize macular pigment distribution in MacTel subjects

DETAILED DESCRIPTION:
One of the earliest manifestations of macular telangiectasia type 2 ("MacTel") is an acquired reduction and/or redistribution of the macular pigment carotenoids at the foveal center. Currently, the biochemical mechanisms and clinical significance underlying these changes are not known, but it seems likely that better understanding of this phenomenon could lead to new interventions against MacTel.

Dr. Bernstein's laboratory at the Moran Eye Center of the University of Utah has focused for the past fifteen years on the role of the macular pigment carotenoids, lutein and zeaxanthin, in maintaining macular health. These xanthophyll carotenoids are derived exclusively from the diet, especially from green leafy vegetables and orange-yellow fruits and vegetables. They are thought to protect the macula from light-induced oxidative damage by virtue of their light-screening and antioxidant properties. Dietary supplement products, from infant formula to those aimed at seniors, primarily contain lutein; however the central macula (the fovea) actually has been shown to have higher concentrations of zeaxanthin.

Dr. Bernstein's lab has identified and characterized the binding proteins responsible for the uptake and stabilization of lutein and zeaxanthin in the macula, developed new, noninvasive methods to quantify and image carotenoids in the retina and many other non-ocular tissues, and has participated in intervention trials of lutein and zeaxanthin against age-related macular degeneration. As a leading site for identification of MacTel families in North America as part of the "MacTel Project", Dr. Bernstein and other researchers at the University of Utah have unique expertise in the biochemistry and biophysics of the macular pigment carotenoids that may help to hasten progress toward effective diagnosis and intervention against MacTel in a highly collaborative manner.

Macular Pigment Imaging:

Dr. Bernstein has extensive experience with various methods to image and quantify macular pigment in the living human eye, especially using autofluorescence imaging (AFI) and resonance Raman imaging (RRI). Dr. Bernstein is also currently utilizing these methods to evaluate age-related macular degeneration (AMD) patients participating in the "AREDS2" study.

The objectives of this study are two-fold:

1. To image the maculas of MacTel subjects using two-wavelength autofluorescence imaging (AFI) and resonance Raman imaging (RRI) to target the 7-degree radius pigment ring characteristic of macular telangiectasia type 2 in order to gain further insight into the significance of this early clinical sign;
2. To evaluate whether supplementation with oral zeaxanthin can normalize macular pigment distribution in MacTel subjects.

This is an open-label pilot study that will enroll up to ten patients affected with macular telangiectasia type 2 and evaluate them every six months for two years. All participants will take 20 mg of zeaxanthin supplement per day for the duration of the study. Macular pigment distributions will be determined using two-wavelength autofluorescence imaging and resonance Raman imaging.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who have MacTel and can conveniently travel to the University of Utah for study evaluations

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to ten subjects of either gender who have MacTel (as confirmed by the MacTel central study Reading Center) will be invited to participate. Only those who can conveniently travel to the University of Utah for study evaluations will be approached since the project does not have sufficient funding to reimburse for travel expenses. Participants must agree to discontinue use of any other supplements containing substantial amounts of carotenoids for one month prior to the baseline visit and for the duration of the study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in macular pigment distribution and concentration | 1 year
  The primary outcome measure will be will be change from baseline in macular pigment distribution and concentration.

SECONDARY OUTCOMES:
Change in visual acuity | 1 year
  Secondary outcome measures will be best-corrected visual acuity, contrast sensitivity, and changes in retinal thickness measured by spectral domain OCT (optical coherence tomography).

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Bernstein, M.D., Ph.D., Principal Investigator — University of Utah
Locations (1):
- Moran Eye Center, University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Bernstein PS, Delori FC, Richer S, van Kuijk FJ, Wenzel AJ. The value of measurement of macular carotenoid pigment optical densities and distributions in age-related macular degeneration and other retinal disorders. Vision Res. 2010 Mar 31;50(7):716-28. doi: 10.1016/j.visres.2009.10.014. Epub 2009 Oct 23. PMID 19854211
- [Background] Bhosale P, Li B, Sharifzadeh M, Gellermann W, Frederick JM, Tsuchida K, Bernstein PS. Purification and partial characterization of a lutein-binding protein from human retina. Biochemistry. 2009 Jun 9;48(22):4798-807. doi: 10.1021/bi9004478. PMID 19402606
- [Background] Sharifzadeh M, Zhao DY, Bernstein PS, Gellermann W. Resonance Raman imaging of macular pigment distributions in the human retina. J Opt Soc Am A Opt Image Sci Vis. 2008 Apr;25(4):947-57. doi: 10.1364/josaa.25.000947. PMID 18382494
- [Background] Loane E, Nolan JM, O'Donovan O, Bhosale P, Bernstein PS, Beatty S. Transport and retinal capture of lutein and zeaxanthin with reference to age-related macular degeneration. Surv Ophthalmol. 2008 Jan-Feb;53(1):68-81. doi: 10.1016/j.survophthal.2007.10.008. PMID 18191658
- [Background] Bhosale P, Bernstein PS. Vertebrate and invertebrate carotenoid-binding proteins. Arch Biochem Biophys. 2007 Feb 15;458(2):121-7. doi: 10.1016/j.abb.2006.10.005. Epub 2006 Oct 30. PMID 17188641
- [Background] Sharifzadeh M, Bernstein PS, Gellermann W. Nonmydriatic fluorescence-based quantitative imaging of human macular pigment distributions. J Opt Soc Am A Opt Image Sci Vis. 2006 Oct;23(10):2373-87. doi: 10.1364/josaa.23.002373. PMID 16985523
- [Background] Bhosale P, Larson AJ, Frederick JM, Southwick K, Thulin CD, Bernstein PS. Identification and characterization of a Pi isoform of glutathione S-transferase (GSTP1) as a zeaxanthin-binding protein in the macula of the human eye. J Biol Chem. 2004 Nov 19;279(47):49447-54. doi: 10.1074/jbc.M405334200. Epub 2004 Sep 7. PMID 15355982
- [Background] Bhosale P, Serban B, Zhao DY, Bernstein PS. Identification and metabolic transformations of carotenoids in ocular tissues of the Japanese quail Coturnix japonica. Biochemistry. 2007 Aug 7;46(31):9050-7. doi: 10.1021/bi700558f. Epub 2007 Jul 14. PMID 17630780